CLINICAL TRIAL: NCT00357968
Title: Protocol H7T-MC-TABL(a) PRasugrel IN Comparison to Clopidogrel for Inhibition of PLatelet Activation and AggrEgation (PRINCIPLE) - TIMI 44
Brief Title: Trial in Subjects Undergoing Cardiac Catheterization With Planned Percutaneous Coronary Intervention With Stenting
Acronym: PRINCIPLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo (Industry); The TIMI Study Group (Other)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10635; H7T-MC-TABL (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Results first posted 2010-08-09 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel to Clopidogrel (Experimental): One time oral loading dose (LD) of 60-mg Prasugrel and placebo matched to clopidogrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by 10-mg Prasugrel and placebo matched to clopidogrel taken orally once a day for 14 days. Patients cross-over to 150 mg clopidogrel and placebo matched to prasugrel taken orally once a day for the next 14 days.
  Interventions: Drug: Prasugrel; Drug: Clopidogrel; Drug: Placebo for Prasugrel; Drug: Placebo for Clopidogrel
- Clopidogrel to Prasugrel (Active Comparator): One time oral LD of 600 mg clopidogrel and placebo matched to prasugrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by 150 mg clopidogrel and placebo matched to prasugrel taken orally once a day for 14 days. Patients cross-over to 10 mg prasugrel and placebo tablets matched to clopidogrel taken orally once a day for the next 14 days.
  Interventions: Drug: Prasugrel; Drug: Clopidogrel; Drug: Placebo for Prasugrel; Drug: Placebo for Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Administered orally
  Other Names: LY 640315; Effient; Efient
Drug: Clopidogrel — Administered orally
Drug: Placebo for Prasugrel — Administered orally
Drug: Placebo for Clopidogrel — Administered orally

SUMMARY:
The purpose of this study is to provide information of the relative potency of prasugrel and clopidogrel on platelet function studies, inflammation, and myocyte necrosis in subjects undergoing elective percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Subjects greater than or equal to 18 years of age undergoing cardiac catheterization with planned percutaneous coronary intervention (if coronary anatomy is suitable) for an indication of chest pain +/or anginal equivalent felt by the treating physician to be related to coronary ischemia.
* At least one of the following (a through c):

  1. Functional study (exercise, or pharmacologic) within the past 8 weeks consistent with ischemia as manifested by at least one of the following:

     1. A reversible defect on nuclear imaging.
     2. A reversible wall-motion abnormality by echocardiography.
     3. Horizontal or down-sloping ST-depressions greater than 1 mm on electrocardiogram (ECG) (if no imaging performed).
  2. Prior coronary revascularization [percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)].
  3. A cardiac catheterization with at least one coronary artery lesion amenable to PCI (not yet performed) within 14 days prior to enrollment.

Exclusion Criteria:

* Known creatine kinase-myocardial bands (CK-MB)or cardiac troponin greater than the upper limit of normal at time of screening
* Planned PCI for acute myocardial infarction (MI) or planned PCI within 48 hours of fibrinolytic therapy for ST segment elevation myocardial infarction (STEMI)
* Have cardiogenic shock at the time of screening (systolic blood pressure 90 mm Hg associated with clinical evidence of end-organ hypoperfusion, or subjects requiring vasopressors to maintain systolic blood pressure over 90 mm Hg and associated with clinical evidence of end-organ hypoperfusion).
* Refractory ventricular arrhythmias
* Have New York Heart Association Class IV congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2006-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rapid City, South Dakota
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Krozingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Giessen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
- Israel (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Prasugrel to Clopidogrel: One time oral loading dose (LD) of 60-mg prasugrel and placebo matched to clopidogrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by a once daily 10-mg prasugrel and placebo matched to clopidogrel (prasugrel maintenance dose) taken orally for 14 days (Treatment 1 Phase). Patients cross-over to a once daily 150-mg clopidogrel and placebo matched to prasugrel (clopidogrel maintenance dose) taken orally for the next 14 days (Treatment 2 Phase).
- Clopidogrel to Prasugrel: One time oral loading dose (LD) of 600-mg clopidogrel and placebo matched to prasugrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by a once daily 150-mg clopidogrel and placebo matched to prasugrel (clopidogrel maintenance dose) taken orally for 14 days (Treatment 1 Phase). Patients cross-over to a once daily 10-mg prasugrel and placebo matched to clopidogrel (prasugrel maintenance dose) taken orally for the next 14 days (Treatment 2 Phase).
Period: First Maintenance Dose Phase
Arm/Group | Prasugrel to Clopidogrel | Clopidogrel to Prasugrel
Started | 102 | 99
Received Loading Dose | 102 | 99
Percutaneous Coronary Intervention (PCI) | 55 | 57
Started Maintenance Dose | 55 | 55
Completed | 54 | 55
Not Completed | 48 | 44
Not completed — Not a PCI patient | 47 | 42
Not completed — Withdrawal by Subject | 1 | 2
Period: Crossover Maintenance Dose Phase
Arm/Group | Prasugrel to Clopidogrel | Clopidogrel to Prasugrel
Started | 54 (1 subject discontinued study drug-did not take clopidogrel during the 2nd phase but completed study) | 55
Completed | 54 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prasugrel to Clopidogrel: One time oral loading dose (LD) of 60-mg prasugrel and placebo matched to clopidogrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by a once daily 10-mg prasugrel and placebo matched to clopidogrel (prasugrel maintenance dose) taken orally for 14 days. Patients cross-over to a once daily 150-mg clopidogrel and placebo matched to prasugrel (clopidogrel maintenance dose) taken orally for the next 14 days.
- Clopidogrel to Prasugrel: One time oral loading dose (LD) of 600-mg clopidogrel and placebo matched to prasugrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by a once daily 150-mg clopidogrel and placebo matched to prasugrel (clopidogrel maintenance dose) for 14 days. Patients cross-over to a once daily 10-mg prasugrel and placebo matched to clopidogrel (prasugrel maintenance dose) taken orally for the next 14 days.
- Total: Total of all reporting groups
Arm/Group | Prasugrel to Clopidogrel | Clopidogrel to Prasugrel | Total
Number analyzed (Participants) | 102 | 99 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 47 | 93
  >=65 years | 56 | 52 | 108
Age Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.73) | 63.8 (9.38) | 63.9 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 22 | 51
  Male | 73 | 77 | 150
Race/Ethnicity, Customized [Number; unit: participants]
  African | 3 | 4 | 7
  Caucasian | 97 | 94 | 191
  Native American | 2 | 0 | 2
  West Asian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  France | 3 | 3 | 6
  Germany | 55 | 53 | 108
  Israel | 15 | 13 | 28
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Inhibition of Platelet Aggregation (IPA) to 20 Micromolar (μM) Adenosine Diphosphate (ADP) at 6 Hours After the Loading Dose
Description: IPA was defined as (1 - [maximal platelet aggregation(MPA) at 6 hours after study drug treatment]/[MPA before drug treatment]) x 100.
Time Frame: 6 hours after loading dose
Population: Consists of all patients who received a loading dose of the study drug, did not receive a glycoprotein (GP) IIb/IIIa antagonist, and had evaluable pre-treatment and 6 hour MPA measurements.
  Patients had received a single loading dose of either 60-mg prasugrel or 600-mg clopidogrel but had not yet received any maintenance dosing.
Measure: Mean (Standard Deviation); unit: percent inhibition
Groups:
- Prasugrel: Patients randomized to a single oral loading dose (LD) of 60-mg prasugrel and placebo matched to clopidogrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended), prior to administration of any maintenance dose.
- Clopidogrel: Patients randomized to a single oral loading dose (LD) of 600-mg clopidogrel and placebo matched to prasugrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended), prior to the administration of any maintenance dose.
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 72 | 77
percent inhibition | 74.81 (13.01) | 31.77 (21.07)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 43.21, 95% CI 2-sided [38.04 to 48.38]

2. Primary Outcome: Inhibition of Platelet Aggregation to 20 μM Adenosine Diphosphate After 14 Days of Maintenance Dose Treatment
Description: Measures IPA during maintenance dosing before and after cross-over for each therapy.
  IPA was defined as (1 - [maximal platelet aggregation(MPA) at 14 days after study drug treatment]/[MPA before drug treatment]) x 100.
Time Frame: after 14 days of maintenance dosing
Population: Includes patients who received a loading dose and underwent percutaneous coronary intervention (PCI) regardless of GP IIb/IIIa antagonist use (this includes subjects who received prasugrel and clopidogrel, in either order, during crossover)
Measure: Mean (Standard Deviation); unit: percent inhibition
Groups:
- Prasugrel: Includes total number of evaluable samples from patients who received prasugrel in each maintenance dose period (40 in the first maintenance period and 45 in the second maintenance period).
- Clopidogrel: Includes total number of evaluable samples from patients who received clopidogrel in each maintenance dose period (46 from the first maintenance dose period and 40 from the second maintenance dose period).
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 85 | 86
percent inhibition | 61.34 (17.84) | 46.06 (21.34)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean difference = 14.93, 95% CI 2-sided [10.6 to 19.26]

3. Secondary Outcome: Inhibition of Platelet Aggregation to 20 μM Adenosine Diphosphate at 2 Hours After the Loading Dose
Description: IPA was defined as (1 - [maximal platelet aggregation (MPA) at 2 hours after study drug treatment]/[MPA before drug treatment]) x 100.
Time Frame: 2 hours after loading dose
Population: Includes all patients who received a loading dose of study drug, did not receive a GP IIb/IIIa antagonist and had evaluable pretreatment and 2 hour MPA measurements. Patients had received a single loading dose of either 60-mg prasugrel or 600-mg clopidogrel but had not yet received any maintenance dosing.
Measure: Mean (Standard Deviation); unit: percent inhibition
Groups:
- Clopidogrel: Patients randomized to a single oral loading dose (LD) of 600-mg clopidogrel and placebo matched to prasugrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended), prior to administration of any maintenance dose.
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 74 | 78
percent inhibition | 64.54 (20.43) | 20.32 (20.22)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 44.75, 95% CI 2-sided [38.35 to 51.15]

4. Secondary Outcome: Number of Participants With Non-Coronary Artery Bypass Graft (CABG) Thrombolysis in Myocardial Infarction (TIMI) Major or Minor Bleeding During the First Maintenance Dose Phase
Description: Non-CABG-related TIMI major bleeding was any intracranial hemorrhage OR any clinically overt bleeding associated with a fall in hemoglobin >=5 gm/dL.
  Non-CABG-related TIMI minor bleeding was any clinically overt bleeding associated with a fall in hemoglobin >=3 gm/dL but <5 gm/dL.
Time Frame: after 14 days of treatment (before cross-over)
Population: Patients received a single loading dose and 14 days of maintenance therapy. Patients had not yet crossed-over to the alternate maintenance dose.
Measure: Number; unit: participants
Groups:
- Prasugrel: Patients randomized to a single oral loading dose (LD) of 60-mg prasugrel and placebo matched to clopidogrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by a 10-mg prasugrel and placebo matched to clopidogrel (prasugrel maintenance dose) taken orally once daily for 14 days.
- Clopidogrel: Patients randomized to a single oral loading dose (LD) of 600-mg clopidogrel and placebo matched to prasugrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by a 150-mg clopidogrel and placebo matched to prasugrel (clopidogrel maintenance dose) taken orally once daily for 14 days.
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 102 | 99
participants | 2 | 0

5. Secondary Outcome: Number of Participants With Non-Coronary Artery Bypass Graft (CABG) Thrombolysis in Myocardial Infarction (TIMI) Major or Minor Bleeding During the Crossover Maintenance Dose Phase
Description: as for outcome 4
Time Frame: 14 days after cross-over
Population: All patients who received a loading dose of study drug, received maintenance therapy for 14 days and then switched to the alternate maintenance therapy.
Measure: Number; unit: participants
Groups:
- Clopidogrel: Patients randomized to a single oral loading dose (LD) of 60-mg prasugrel and placebo matched to clopidogrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by a 10-mg prasugrel prasugrel and placebo matched to clopidogrel (prasugrel maintenance dose) taken orally once daily for 14 days. Patients crossed over to a 150-mg clopidogrel and placebo matched to prasugrel (clopidogrel maintenance dose) taken orally for the next 14 days.
- Prasugrel: Patients randomized to a single oral loading dose (LD) of 600-mg clopidogrel and placebo matched to prasugrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by a 150-mg clopidogrel and placebo matched to prasugrel (clopidogrel maintenance dose) taken orally once daily for 14 days. Patients crossed over to a 10-mg prasugrel and placebo matched to clopidogrel (prasugrel maintenance dose) taken orally for the next 14 days.
Arm/Group | Clopidogrel | Prasugrel
Number analyzed (Participants) | 53 | 55
participants | 0 | 0

6. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE) During the First Maintenance Dose Phase
Description: Number of patients who met any of the following endpoints: cardiovascular death, myocardial infarction, stroke, subacute stent thrombosis, or urgent target vessel revascularization
Time Frame: after 14 days of treatment (before cross-over)
Population: Includes all patients who received a loading dose. Patients who underwent PCI also received 14 days of maintenance treatment. Patients had not yet crossed-over to the alternate maintenance treatment.
Measure: Number; unit: participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 102 | 99
participants | 2 | 1

7. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events During the Crossover Maintenance Dose Phase
Description: as for outcome 6
Time Frame: 14 days after cross-over
Population: Includes all patients who received a loading dose and underwent PCI, received a maintenance dose for 14 days, and then crossed-over to the alternate therapy for an additional 14 days of maintenance dosing.
Measure: Number; unit: participants
Groups:
- Clopidogrel: Patients randomized to a single oral loading dose (LD) of 60-mg prasugrel and placebo matched to clopidogrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by a 10-mg prasugrel and placebo matched to clopidogrel (prasugrel maintenance dose) taken orally once daily for 14 days. Patients crossed over to a 150-mg clopidogrel and placebo matched to prasugrel (clopidogrel maintenance dose) for the next 14 days.
- Prasugrel: Patients randomized to a single oral loading dose (LD) of 600-mg clopidogrel and placebo matched to prasugrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by a 150-mg clopidogrel and placebo matched to prasugrel (clopidogrel maintenance dose) taken orally once daily for 14 days. Patients crossed over to a 10-mg prasugrel and placebo matched to clopidogrel (prasugrel maintenance dose) for the next 14 days.
Arm/Group | Clopidogrel | Prasugrel
Number analyzed (Participants) | 53 | 55
participants | 1 | 0

8. Secondary Outcome: Number of Hyporesponsive Participants at 6 Hours After the Loading Dose
Description: Number of patients with inhibition of platelet aggregation (IPA) with 20 uM adenosine diphosphate (ADP) <20%
Time Frame: 6 hours after loading dose
Population: Includes patients who received a loading dose of the study drug, did not receive a glycoprotein (GP) IIb/IIIa antagonist and had evaluable pre-treatment, and 6 hour MPA measurements.
  Patients had received a single loading dose of either 60-mg prasugrel or 600-mg clopidogrel but had not yet received any maintenance dosing.
Measure: Number; unit: participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 72 | 77
participants | 0 | 21
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.0001, Chi-squared

9. Secondary Outcome: Number of Hyporesponsive Participants at the End of the First Maintenance Dose Phase
Description: Number of patients with inhibition of platelet aggregation (IPA) with 20 uM adenosine diphosphate (ADP) <20%
Time Frame: From loading dose to day 15
Population: Includes patients who received a single loading dose and had evaluable MPA measures, regardless of glycoprotein (GP) IIb/IIIa antagonist use. Patients had received 14 days of maintenance treatment but had not crossed-over to the alternate maintenance treatment.
Measure: Number; unit: participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 40 | 46
participants | 1 | 7
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p = 0.0629, Fisher Exact

10. Secondary Outcome: Number of Hyporesponsive Participants at the End of the Crossover Maintenance Dose Phase
Description: Number of patients with inhibition of platelet aggregation (IPA) with 20 uM adenosine diphosphate (ADP) <20%
Time Frame: 14 days after cross-over
Population: Includes patients who received a single loading dose and had evaluable MPA measures,regardless of glycoprotein (GP) IIb/IIIa antagonist use. Patients received 14 days of maintenance treatment and then crossed-over to the alternate maintenance treatment for 14 days.
Measure: Number; unit: participants
Arm/Group | Clopidogrel | Prasugrel
Number analyzed (Participants) | 40 | 45
participants | 4 | 1
Statistical Analysis 1: Comparison: Clopidogrel vs Prasugrel; Test type: Superiority or Other; p = 0.1827, Fisher Exact

11. Secondary Outcome: Platelet Reactivity Index Percent (PRI%) Measured by Vasodilator-stimulated Phosphoprotein (VASP) at 2 Hours After the Loading Dose
Description: VASP phosphorylation in response to prostaglandin E1 (PGE1) with and without ADP was determined by whole-blood flow cytometry and was expressed as a platelet reactivity index (PRI). PRI was defined as [(MFI(with PGE1) - MFI (with PGE1 and ADP))/MFI(with PGE1) x 100] where MFI is mean fluorescence index. A lower PRI indicates greater antiplatelet effect.
Time Frame: 2 hours after loading dose
Population: Includes patients who received a loading dose, underwent PCI, did not receive a GP IIb/IIIa antagonist, and had evaluable VASP measurements. Patients had received a single loading dose but had not yet received any maintenance treatment.
Measure: Mean (Standard Deviation); unit: percent (%) platelet reactivity index
Groups:
- Clopidogrel: Patients randomized to a single oral loading dose (LD) of 600-mg clopidogrel and placebo matched to prasugrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) prior to any maintenance dose.
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 93 | 88
percent (%) platelet reactivity index | 21.5 (27.06) | 75.0 (16.91)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -54.3, 95% CI 2-sided [-61.2 to -47.4]

12. Secondary Outcome: Platelet Reactivity Index Percent (PRI%) Measured by Vasodilator-stimulated Phosphoprotein (VASP) at 6 Hours After the Loading Dose
Description: as for outcome 11
Time Frame: 6 hours after loading dose
Population: Includes patients who received a loading dose, underwent PCI, and had evaluable VASP measurements, and did not receive a GP IIb/IIIa antagonist. Patients had received a single loading dose but had not yet received any maintenance treatment.
Measure: Mean (Standard Deviation); unit: percent (%) platelet reactivity index
Groups:
- Prasugrel: Patients randomized to a single oral loading dose (LD) of 60-mg prasugrel and placebo matched to clopidogrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) prior to any maintenance dose
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 68 | 68
percent (%) platelet reactivity index | 7.4 (16.66) | 68.4 (21.18)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -60.5, 95% CI 2-sided [-67.1 to -54.0]

13. Secondary Outcome: Platelet Reactivity Index Percent (PRI%) Measured by Vasodilator-stimulated Phosphoprotein (VASP) 18 to 24 Hours After the Loading Dose
Description: VASP phosphorylation in response to prostaglandin E1 (PGE1) with and without ADP was determined by whole-blood flow cytometry and was expressed as a platelet reactivity index (PRI). PRI was defined as [(MFI(with PGE1) - MFI (with PGE1 and ADP))/MFI(with PGE1) x 100] where MFI is mean flourescence index. A lower PRI indicates greater antiplatelet effect.
Time Frame: 18 to 24 hours after loading dose
Population: Includes patients who received a loading dose, underwent PCI, did not receive a GP IIb/IIIa antagonist, and had evaluable VASP measurements.
Measure: Mean (Standard Deviation); unit: percent (%) platelet reactivity index
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 48 | 54
percent (%) platelet reactivity index | 10.3 (15.63) | 64.3 (18.72)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -56.2, 95% CI 2-sided [-63.2 to -49.2]

14. Secondary Outcome: Platelet Reactivity Index Percent (PRI%) Measured by Vasodilator-stimulated Phosphoprotein (VASP) After 14 Days of Maintenance Dose Treatment
Description: as for outcome 11
Time Frame: after 14 days of maintenance dosing
Population: Includes patients who received a loading dose and PCI, regardless of GP IIb/IIIa antagonist use (this includes subjects who received prasugrel and clopidogrel, in either order, during crossover)
Measure: Mean (Standard Deviation); unit: percent (%) platelet reactivity index
Groups:
- Prasugrel: Includes the total number of evaluable samples from patients who received prasugrel in each maintenance dose period (50 from the first maintenance dose period and 50 from the second maintenance dose period)
- Clopidogrel: Includes total number of evaluable samples from patients who received clopidogrel in each maintenance dose period (52 from the first maintenance dose period and 51 from the second maintenance dose period).
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 100 | 103
percent (%) platelet reactivity index | 23.4 (19.19) | 43.8 (23.26)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean difference = -20.1, 95% CI 2-sided [-25.7 to -14.5]

15. Secondary Outcome: Myonecrosis Measure: Creatine Kinase-Myocardial Bands (CK-MB) at 6 Hours After the Loading Dose
Description: Mean CK-MB at 6 hours after loading dose. CK-MB is a biomarker for myonecrosis
Time Frame: 6 hours after loading dose
Population: Includes patients who received a loading dose, underwent PCI, did not receive a GP IIb/IIIa antagonist, and had an evaluable CK-MB measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 45 | 51
IU/L | 9.16 (8.3) | 8.13 (5.16)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p = 0.7058, ANCOVA; Mean Difference (Net) = -0.47, 95% CI 2-sided [-2.95 to 2.00]

16. Secondary Outcome: Myonecrosis Measure: Creatine Kinase-Myocardial Bands (CK-MB) 18 to 24 Hours After the Loading Dose
Description: Mean CK-MB at 18-24 hours after loading dose. CK-MB is a biomarker for myonecrosis.
Time Frame: 18 to 24 hours after loading dose
Population: as for outcome 15
Measure: Median (Standard Deviation); unit: IU/L
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 47 | 51
IU/L | 11.64 (8.22) | 11.16 (8.72)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p = 0.4029, ANCOVA; Mean Difference (Net) = -1.33, 95% CI 2-sided [-4.48 to 1.82]

17. Secondary Outcome: Myonecrosis Measure: Cardiac Troponin at 6 Hours After the Loading Dose
Description: Mean troponin level at 6 hours after the loading dose. Troponin is a biomarker for myonecrosis.
Time Frame: 6 hours after loading dose
Population: Includes patients who received a loading dose, underwent PCI, did not receive a GP IIb/IIIa antagonist, and had an evaluable troponin measure.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 46 | 50
ng/ml | 0.06 (0.204) | 0.05 (0.128)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p = 0.7893, ANCOVA; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.06 to 0.08]

18. Secondary Outcome: Myonecrosis Measure: Cardiac Troponin 18 to 24 Hours After the Loading Dose
Description: Mean troponin level at 18 to 24 hours after the loading dose. Troponin is a biomarker for myonecrosis.
Time Frame: 18 to 24 hours after loading dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 44 | 49
ng/ml | 0.12 (0.273) | 0.13 (0.277)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p = 0.4528, ANCOVA; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.25 to 0.07]

ADVERSE EVENTS:
Groups:
- Prasugrel Before Cross-over: One time oral loading dose (LD) of 60 mg prasugrel and placebo matched to clopidogrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by prasugrel 10 mg and placebo matched to clopidogrel (prasugrel maintenance dose) once daily for 14 days.
- Clopidogrel Before Cross-over: One time oral loading dose of 600 mg clopidogrel and placebo matched to prasugrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by 150 mg clopidogrel and placebo matched to prasugrel (clopidogrel maintenance dose) once daily for 14 days.
- Prasugrel After Cross-over: Prasugrel 10 mg and placebo matched to clopidogrel (prasugrel maintenance dose)once daily for 14 days after cross-over from one time loading dose of clopidogrel 600 mg and placebo matched to prasugrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by clopidogrel 150 mg and placebo matched to prasugrel (clopidogrel maintenance dose) once daily for 14 days
- Clopidogrel After Cross-over: Clopidogrel 150 mg and placebo matched to prasugrel (clopidogrel maintenance dose) once daily for 14 days after cross-over from one time loading dose of 60 mg prasugrel and placebo matched to clopidogrel (plus oral enteric coated aspirin 325 mg to 500 mg is recommended) followed by 10 mg prasugrel and placebo matched to clopidogrel (prasugrel maintenance dose) once daily for 14 days.
Arm/Group | Prasugrel Before Cross-over | Clopidogrel Before Cross-over | Prasugrel After Cross-over | Clopidogrel After Cross-over
Serious Adverse Events (participants affected / at risk) | 8/102 | 7/99 | 1/55 | 3/53
Other Adverse Events (participants affected / at risk) | 40/102 | 40/99 | 16/55 | 12/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel Before Cross-over (N=102) | Clopidogrel Before Cross-over (N=99) | Prasugrel After Cross-over (N=55) | Clopidogrel After Cross-over (N=53)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Borrelia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonmary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIth nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel Before Cross-over (N=102) | Clopidogrel Before Cross-over (N=99) | Prasugrel After Cross-over (N=55) | Clopidogrel After Cross-over (N=53)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 2 (2) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure orthostatic (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac enzymes increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site discharge (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 4 (4) | 3 (3) | 2 (2) | 2 (2)
Coagulation time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Reproductive system and breast disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site complications (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratiry tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Middle insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days